CLINICAL TRIAL: NCT02841566
Title: GAMbling and MAterialism
Brief Title: Comparative Study of the Link Between the Practice of Gambling and Money and Materialism Among Problem Gamblers and Non-problem Gamblers
Acronym: GAMMA
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC15_0372
Record Dates: First submitted 2016-07-19; First posted 2016-07-22 (Estimated); Last update posted 2016-07-22 (Estimated); Status verified 2016-07

CONDITIONS: Gambling
MeSH Terms: conditions — Gambling | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Problem glambers: The group of problem gamblers will consist of patients already included in the cohort EVALADD [favorable opinion of GNEDS 06/09/2012; CNIL authorization No. 912631 of 10.09.2013], and the data will be extracted directly from the database EVALADD
  Interventions: Other: questionnaire
- Non-problem gamblers: The subjects of this group will be matched on sex, age and education level with the group problem gamblers. They will be recruited over the Internet and using the volunteer base [normal declaration with the CNIL: No. 1761543 of 21/05/2014].
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire

SUMMARY:
The purpose of this study is to to explore the link between materialism and addiction to gambling and money

ELIGIBILITY:
Inclusion Criteria: ( specific to problem gamblers)

* subject having at least four diagnostic criteria in "Trouble linked to gambling and money" DSM-5 (APA 2013)
* subject who had written consent for participation in the EVALADD cohort
* Subject who has started treatment for a problem with the practice of gambling and money in the addictology and psychiatric department

( specific to non-problem gamblers)

* Subject playing games of chance and money at least once a year
* Subject playing games of chance and money less than once per week OR less than € 500 per year
* Subject having a score of 0-2 at ICJE questionnaire

Exclusion Criteria:

* Subject having difficulty reading or writing of the French language
* Subject having Parkinson's Disease
* Subject under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All new patients be seen by a doctor for a behavioral addiction in the addictology and psychiatric department
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2015-10; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Materialism level among problem gamblers compared to non-problem gamblers | 1 year
  To assess the total score of materialism by the Material Value Scale in 15 items (MVS-15), among a group of non-problem gamblers and a group of problem gamblers.